CLINICAL TRIAL: NCT01622127
Title: Efficacy of Self-fixating Mesh in Ventral and Incisional Hernia Repair
Brief Title: Progrip Ventral Study for Sublay Repair
Status: Completed | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Collaborators: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Other Study IDs: 2011/497
Record Dates: First submitted 2012-06-14; First posted 2012-06-18 (Estimated); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Primary Ventral and Incisional Hernia Repair

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- incisional hernias
  Interventions: Device: Parietex ProGrip™

INTERVENTIONS:
Device: Parietex ProGrip™ — ProGrip™ mesh is a lightweight (40g/m2) monofilament polypropylene or polyester mesh with resorbable polylactic acid (PLA) micro-grips, which provide self-gripping properties during the first few months after implantation.

SUMMARY:
A novel concept of self-gripping mesh has been developed to achieve secure and long-term posterior wall reinforcement. ProGrip™ mesh is a lightweight (40g/m2) monofilament polypropylene or polyester mesh with resorbable polylactic acid (PLA) micro-grips, which provide self-gripping properties during the first few months after implantation. The self-fixation of the mesh to the underlying tissues is instantly achieved at application, limiting or avoiding the requirement of sutures (which can penetrate underlying tissues and damage cutaneous nerves), and providing a near tension-¬free repair.

Case series confirmed that Parietex ProGrip™ placed in onlay position allows a safe and painless treatment of incisional hernias and provides secure and efficient fixation mesh. On this basis, larger sizes Parietex ProGrip™ meshes have been developed for larger incisional hernia defect treatment. In order to assess the clinical outcomes following the use of ProGrip™ larger sizes in incisional hernia repair, this mono-center observational study has been initiated.

ELIGIBILITY:
Inclusion Criteria:

* All patients at participating hospital undergoing incisional hernia repair by using retromuscular placement by open approach.
* Defect size: 5cm ≤ width*, 10 cm ≤ length ≤ 20 cm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with primary ventral and incisional hernia repair.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2012-02 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Incidence of peri-operative and post-operative complications using Parietex ProGrip™. | 24 months after surgery
  Clinical observation: recurrence, wound complications pain, pain/ chronic pain and other postoperative complications

SECONDARY OUTCOMES:
Description and assessment of the use of Parietex™ ProGrip™ larger sizes meshes at time of surgery | End of surgical procedure

CONTACTS AND LOCATIONS:
Overall Officials: Frederik Berrevoet, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Related Info — http://www.uzgent.be